CLINICAL TRIAL: NCT03002519
Title: A Phase I Open-label Dose-escalation Study to Evaluate the Safety of Intramuscular Injections of PLX-R18 in Subjects With Incomplete Hematopoietic Recovery Following Hematopoietic Cell Transplantation
Brief Title: Safety Evaluation of Intramuscular Injections of PLX-R18 in Subjects With Incomplete Hematopoietic Recovery Following Hematopoietic Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pluristem Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX-R18-HCT-01
Record Dates: First submitted 2016-12-13; First posted 2016-12-23 (Estimated); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Incomplete HCT (Hematopoietic Cell Transplantation)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PLX-R18 (Experimental): Dose Escalation- first three subjects will be enrolled in the low dose cohort, 6 subjects in the intermediate-dose cohort, and 15 subjects in the high dose cohort.
  Interventions: Biological: PLX-R18

INTERVENTIONS:
Biological: PLX-R18 — Intramuscular (IM) administration of PLX-R18

SUMMARY:
This study aims to evaluate the safety of intramuscular (IM) administration of PLX-R18 in subjects with incomplete hematopoietic recovery following HCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. At least 3 months after HCT, either autologous or allogeneic (of any source, with any preparatory regimen, for any indication), prior to study treatment.
3. Sustained platelet count ≤50,000/µL, and/or sustained Hb ≤8 g/dL and/or sustained ANC ≤1000/mm3, attributed to graft failure as a major contributor, as evident by hypocellular bone marrow.

   Cytopenia should be confirmed by at least 2 consecutive blood counts, at least one of them within 28 days prior to treatment (higher transient levels following occasional blood product transfusions are allowed).
4. Stable donor cell chimerism in at least 3 consecutive tests prior to treatment (the most recent test should be within 28 days prior to treatment).
5. If the subject had allogeneic HCT for a malignant disease, the subject should have complete donor chimerism.

   *complete donor chimerism should be determined by the investigator per site's standards.
6. General performance status evaluated by Eastern Cooperative Oncology Group 0-2 scale.
7. Signed written informed consent.

Exclusion Criteria:

INCLUSION AND EXCLUSION CRITERIA Inclusion Criteria

Subjects must meet all of the inclusion criteria listed below to be eligible for the study:

1. Age ≥18 years.
2. At least 3 months after HCT, either autologous or allogeneic (of any source, with any preparatory regimen, for any indication), prior to study treatment.
3. Sustained platelet count ≤50,000/µL, and/or sustained Hb ≤8 g/dL and/or sustained ANC ≤1000/mm3, attributed to graft failure as a major contributor, as evident by hypocellular bone marrow.

Cytopenia should be confirmed by at least 2 consecutive blood counts, at least one of them within 28 days prior to treatment (higher transient levels following occasional blood product transfusions are allowed).

4. Stable donor cell chimerism in at least 3 consecutive tests prior to treatment (the most recent test should be within 28 days prior to treatment).

5. If the subject had allogeneic HCT for a malignant disease, the subject should have complete donor chimerism.

*complete donor chimerism should be determined by the investigator per site's standards.

6. General performance status evaluated by Eastern Cooperative Oncology Group 0-2 scale.

7. Signed written informed consent. Exclusion Criteria

1. Evidence of developing malignancy since the HCT, or any evidence of malignancy at the time of screening.
2. Current active infection requiring systemic treatment (if infection resolved but antibiotic coverage continues, patient may be included).
3. Acute graft versus host disease (GvHD) Grade III or IV, or severe chronic GvHD at the time of screening.
4. Subject has received prophylactic treatment with donor lymphocyte infusion (DLI) within 6 months prior to treatment, or any other cell therapy within 3 months prior to treatment.
5. History of malignancy (other than the disease that required the HCT) within 2 years prior to screening (except for skin basal cell carcinoma or squamous cell carcinoma lesions that were fully resected with no need for further treatment, and not located at the injection site).
6. History of significant transfusion reaction including: Transfusion related acute lung injury (pulmonary edema), shock, severe disturbances of liver function tests, renal dysfunction, or hemolytic anemia (as part of the transfusion reaction).
7. Known allergies to any of the following: dimethyl sulfoxide (DMSO), human serum albumin, bovine serum albumin, gentamicin, or antihistamine.
8. History of allergic/hypersensitivity reaction to any substance having required hospitalization and/or treatment with intra-venous steroids/epinephrine or in the opinion of the Investigator the subject is at high risk of developing severe allergic/hypersensitivity reactions (does not apply to transfusion reactions - see exclusion criterion 8).
9. A known history of allergic/hypersensitivity reactions to 3 or more allergens.
10. History of uncontrolled asthma (Global Initiative for Asthma Grade III IV).
11. History of severe atopic disease (including but not limited to chronic urticaria, allergic reaction with respiratory symptoms requiring systemic steroids).
12. Medical history of human immunodeficiency virus or syphilis infection.
13. Known active hepatitis B or hepatitis C infection at the time of screening.
14. A pregnant or lactating woman or a woman who plans to become pregnant during the study. In addition, any woman of childbearing potential (not sterile or postmenopausal), who is unwilling to adhere to the use of a highly effective contraception method for the duration of the study:

    1. Oral/intravaginal/transdermal combined estrogen and progestogen containing hormonal contraception for at least 3 months prior to screening.
    2. Oral/injectable/implantable progestogen-only hormonal contraception for at least 3 months prior to screening.
    3. An intrauterine device (IUD) or intrauterine hormone-releasing system (IUS).
15. Subjects on renal replacement therapy or with estimated glomerular filtration rate (eGFR) <15 mL/min/1.73m2 (based on Modification of Diet in Renal Disease [MDRD] equation).
16. Serum glutamic pyruvic transaminase (alanine aminotransferase), serum oxaloacetic pyruvic transaminase (aspartate aminotransferase) >2.5 x upper limit of normal range.
17. International normalized ratio (INR) >2 or subjects who are on oral anticoagulant therapy with INR >2 unless anticoagulation treatment can be safely interrupted/discontinued around each investigational product (IP) treatment upon primary care physician and/or Investigator's discretion.
18. Severe or uncontrolled/unstable cardiac, pulmonary, or renal disease, including myocardial infarction or cerebrovascular accident within 3 months prior to treatment.
19. History of solid organ transplantation.
20. Signs and symptoms of active central nervous system disease.
21. Life expectancy <6 months as assessed by the Investigator.
22. Subject has participated in a clinical interventional study and received the last treatment within 30 days prior to screening.
23. In the opinion of the Investigator, the subject is unsuitable for participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Emergent Adverse Events (AEs) | Recorded after time of consent throughout the study until the last visit (~1 year)
Safety laboratory values (including immunological testing) | Blood samples will be collected on each visit, through study completion (~1 year)
Vital signs | Will be assessed during each visit, through study completion (~1 year)
ECG | Will be assessed during the screening visit, before each IP treatment visit and on the 14th day of participation (visit 5).

CONTACTS AND LOCATIONS:
Locations (10):
- United States (7):
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Kansas Cancer Center - The Richard and Annette Bloch Cancer Care Pavilion,2330 Shawnee Mission Parkway, Westwood, Kansas
  - University of Maryland Medical Center,22 South Greene Street, Baltimore, Maryland
  - Mayo Clinic Cancer Center (MCCC) - Rochester,200 1st Street SW, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Baylor University Medical Center, Dallas, Texas
- Israel (3):
  - Rambam Medical Center, Haifa
  - Hadassah Ein Karem Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan

REFERENCES:
- [Derived] McGuirk JP, Metheny L 3rd, Pineiro L, Litzow M, Rowley SD, Avni B, Tamari R, Lazarus HM, Rowe JM, Sheleg M, Rothenstein D, Halevy N, Zuckerman T. Placental expanded mesenchymal-like cells (PLX-R18) for poor graft function after hematopoietic cell transplantation: A phase I study. Bone Marrow Transplant. 2023 Nov;58(11):1189-1196. doi: 10.1038/s41409-023-02068-3. Epub 2023 Aug 8. PMID 37553467